CLINICAL TRIAL: NCT03319407
Title: EPAD Monitoring of Patients Undergoing Robotic Assisted Laparoscopic Genitourinary Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding support unavailable
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert McClain, MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-006546
Record Dates: First submitted 2017-10-20; First posted 2017-10-24 (Actual); Results first posted 2019-10-30 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Observation (Other): All participants will be monitored with EPAD system
  Interventions: Device: EPAD monitoring system

INTERVENTIONS:
Device: EPAD monitoring system — EPAD system will be used as part of routine care

SUMMARY:
Participants to be enrolled in this study will have been scheduled to have laparoscopic genitourinary surgery and EPAD monitoring as part of their clinical care intraoperatively. Patients scheduled for genitourinary surgery are often at risk for developing nerve injuries due to intraoperative positioning.

Somatosensory evoked potential devices (SSEP) are commonly used to detect pending injury to peripheral nerves. The purpose of the present study is to use SSEP monitoring to determine the incidence and potential causes of significant changes in SSEP waveforms and correlate these changes with neurologic status of the brachial plexus after robotic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo robotic assisted laparoscopic genitourinary surgery
* Patients who are scheduled to have EPAD monitoring as part of their clinical care intraoperatively

Exclusion Criteria:

• Patients with previous history of polyneuropathy, carpal tunnel, ulnar neuropathy, or similar neurological deficiencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert McClain, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observation
Started | 21
Completed | 0
Not Completed | 21

BASELINE CHARACTERISTICS:
Arm/Group | Observation
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Somatosensory Evoked Potential Monitoring
Description: Recording of somatosensory evoked potential in patients undergoing genitourinary surgery
Time Frame: in the first 24 hours of postoperative period
Population: Study terminated prematurely. Data was not collected.
Arm/Group | Observation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over a 24 hour period.
Arm/Group | Observation
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT03319407/Prot_SAP_000.pdf